CLINICAL TRIAL: NCT05119218
Title: Gut Microbiota Profile, SCFA, Gut Integrity, Parasite Infection, Hygiene Practice and Cognitive Score on Stunted Children in East Nusa Tenggara
Brief Title: Gut Microbiota Stunted Children NTT
Status: Completed | Type: Observational
Sponsor: Bina Nusantara University (Other)
Collaborators: Kementerian Riset dan Teknologi / Badan Riset dan Inovasi Nasional, Indonesia (Other Government); Maastricht University (Other); Universitas Airlangga (Other); Yarsi University (Unknown); Universitas Kristen Indonesia (Other)
Responsible Party: Principal Investigator, Ingrid S Surono, Principal Investigator, Bina Nusantara University
Other Study IDs: 332/KEP-UY/BIA/X/2021
Record Dates: First submitted 2021-11-02; First posted 2021-11-15 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Stunting
Keywords: stunting; Gut microbiota; toddler; SCFA; Parasite; Hygiene Practice
MeSH Terms: conditions — Growth Disorders

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Biospecimen Retention: Samples With DNA — stool and blood sampling
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stunted subject: The population is all children under five aged 3-5 years in the stunting locus village. Subjects in this study were taken with a sampling quota of 100 stunting toddlers toddlers in each area.
  Interventions: Other: No Intervention
- Normal subject: The population is all children under five aged 3-5 years in the stunting locus village. Subjects in this study were taken with a sampling quota of 100 non-stunted toddlers in each area.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
NTT Province is on the list of priority areas of high prevalence of stunting, Southwest Sumba, South Middle East, and Kupang district have a stunting prevalence of 36.2%, 34.5% and 48.1% respectively in 2020. Therefore, it is necessary to conduct a profile study. microbiota, SCFA, gastrointestinal integrity, parasites, hygiene practice, and cognition in stunting and healthy toddlers in the province of East Nusa Tenggara,

DETAILED DESCRIPTION:
Stunting indicates a public health problem because it is associated with an increased risk of morbidity and mortality, decreased motor and mental function development, and reduced physical capacity. Stunting is a chronic nutritional deficiency condition that affects the growth and development, and intelligence of children. Lack of nutrients can cause intestinal microbiota dysbiosis where this will reduce the metabolism of short chain fatty acids (SCFA) which will affect the absorption of nutrients in the small intestine and cause impaired immunity, which in turn worsens stunting conditions. The composition of the gut microbiota is influenced by age, sex, geographic area and food intake. Therefore, the description of knowledge, attitudes and applications in society, especially mothers and child subjects, was also analyzed using a hygiene practice questionnaire. The aim of the study was to obtain an overview of the gut microbiota, gastrointestinal integrity, parasitic infections, hygiene practices and cognitive scores in stunting and healthy toddlers in several areas in the province of East Nusa Tenggara as a baseline study to be followed up by intervention study.

The research will be conducted for 3 (three) months in 2021/2022. The subjects involved represented 100 stunted children and 100 healthy children aged 36-45 months from each region. Determination of the sample with a sampling quota. The variables studied were the nutritional status of under five years children, characteristics of children under five (age, gender, birth weight (BBL), birth length, breast feeding history, immunization history, history of diarrhea, history of ARI (Upper Respiratory Tract Infection)), mother and family characteristics (age, education). , occupation, father's occupation, total family income), home environment and hygiene, vaccination history, gastrointestinal microbiota status, gastrointestinal integrity, parasites, hygiene practices, and cognitive scores.

ELIGIBILITY:
Inclusion Criteria:

* Anthropometric measurements of stunting were measured based on the parameters of length/height according to age compared to the 2005 WHO anthropometric standards and the Indonesian Ministry of Health Decree No. 1995/MENKES/SK/XII/2010.

Exclusion Criteria:

* criteria thats makes subject appropiate, like more than 5 years old, not live in sampling area, unhealthy

Ages: 36 Months to 45 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This observational study used a cross sectional design with a quantitative approach. The cross-sectional research design is a research conducted at one time and one time to find the relationship between the independent variable (risk factor) and the dependent variable (effect) as baseline data
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-02-20 (Actual)

PRIMARY OUTCOMES:
200 sample Gut Microbiota Profile descript OTU by NGS | 2 months
  Profile of genus microbiota observed using Next Generation Sequencing

SECONDARY OUTCOMES:
200 sample Short Chain Fatty Acid Profile from feses sample | 1 months
  microbiota metabolite profile
200 sample Gut Integrity profile from blood sample | 2 months
  serum lipid binding protein, serum citrulline, serum Intestinal Fatty Acid Binding Protein (IFABP), serum Fatty Acid Binding Protein (FABP), sCD14, dan sCD163.
200 sample immune response from blood sample | 2 months
  TNF, TGF, IL-10, dan sIgA
200 data hygiene practice from quenstionare data | 2 months
  epidemiology data, daily hygiene practice, family data
200 cognitive development data from coqnitive measurement | 2 months
  coqnitive descriptive

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid S Surono, PhD, Principal Investigator — Bina Nusantara University
Locations (1):
- University, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No
planned not to be shared

REFERENCES:
- [Background] Surono IS, Jalal F, Bahri S, Romulo A, Kusumo PD, Manalu E, Yusnita, Venema K. Differences in immune status and fecal SCFA between Indonesian stunted children and children with normal nutritional status. PLoS One. 2021 Jul 29;16(7):e0254300. doi: 10.1371/journal.pone.0254300. eCollection 2021. PMID 34324500
- [Result] Surono IS, Widiyanti D, Kusumo PD, Venema K. Gut microbiota profile of Indonesian stunted children and children with normal nutritional status. PLoS One. 2021 Jan 26;16(1):e0245399. doi: 10.1371/journal.pone.0245399. eCollection 2021. PMID 33497390
- [Derived] Surono IS, Athiyyah AF, Venema K. Gut microbiota, SCFA and nutritional intake in stunted children in East Nusa Tenggara, Indonesia. Benef Microbes. 2025 Jul 24;16(6):647-658. doi: 10.1163/18762891-bja00090. PMID 40716760
- [Derived] Surono IS, Popov I, Verbruggen S, Verhoeven J, Kusumo PD, Venema K. Gut microbiota differences in stunted and normal-lenght children aged 36-45 months in East Nusa Tenggara, Indonesia. PLoS One. 2024 Mar 29;19(3):e0299349. doi: 10.1371/journal.pone.0299349. eCollection 2024. PMID 38551926